CLINICAL TRIAL: NCT02863679
Title: Topical Anesthesia of Tetracaine Hydrochloride Jelly on Cervix After Hysteroscopic Uterine Stent Insertion
Brief Title: Postoperative Analgesic Efficacy of Tetracaine Hydrochloride Gel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Feng Lin, attending doctor, Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tetracaine hydrochloride gel
Record Dates: First submitted 2016-08-08; First posted 2016-08-11 (Estimated); Last update posted 2016-10-12 (Estimated); Status verified 2016-10

CONDITIONS: Hysteroscopy
Keywords: tetracaine hydrochloride gel; analgesia; intrauterine balloon; hysteroscope operation
MeSH Terms: conditions — Agnosia | interventions — Tetracaine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tetracaine hydrochloride gel group (Experimental): Patients in getracaine hydrochloride gel group were covered with a gauze with tetracaine hydrochloride gel on the cervix after hysteroscopic insertion of utrauterine balloon stent.
  Interventions: Drug: Tetracaine hydrochloride gel
- Control group (Placebo Comparator): Patients in control group were covered with a gauze with saline on the cervix after hysteroscopic insertion of utrauterine balloon stent.
  Interventions: Drug: Tetracaine hydrochloride gel

INTERVENTIONS:
Drug: Tetracaine hydrochloride gel — Tetracaine hydrochloride gel contains 1% tetracaine hydrochloride, and a fair dose of fungicide, lubricants, remove foam agent, as the long-term local anesthetics.
  Other Names: Tetracaine HCL

SUMMARY:
This study was taken out to assess the postoperative analgesic efficacy of tetracaine hydrochloride gel in patients with intrauterine adhesion treating with intrauterine balloon.Participates were assigned into two groups by randomly-tetracaine hydrochloride gel group and control group.

DETAILED DESCRIPTION:
Tetracaine hydrochloride gel contains 1% tetracaine hydrochloride, and a fair dose of fungicide, lubricants, remove foam agent, as the long-term local anesthetics. Patients in getracaine hydrochloride gel group were covered with a gauze of tetracaine hydrochloride gel on the external cervical orifice after insert an utrauterine balloon in the uterine cavity. While patients in the control group were covered with a blank gauze after hysteroscopic adhesiolysis. Compare the postoperative analgesic scor and patients' analgesic satisfaction of the two groups and asess the analgesic efficacy of tetracaine hydrochloride gel.

ELIGIBILITY:
Inclusion Criteria:

* no previous history of hysteroscopic adhesiolysis or surgery on the cervix
* inserted intrauterine balloon in the uterine cavity after hysteroscopic adhesiolysis
* no other diseases

Exclusion Criteria:

* Allergy to local anesthetics
* Patients with chronic pain
* Patients with abnormal blood coagulation function
* Patients with mental illness that can not cooperate
* Patients with previous hysteroscopic adhesiolysis or cervical surgery

Ages: 19 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Numerical Rating Scale (NRS) score | 7 days

SECONDARY OUTCOMES:
patients received balloon volume reduction | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Feng Lin, MD, Principal Investigator — The 1st Affiliated Hospital of Wenzhou Medical University
Locations (1):
- the 1st Affiliated Hospital of Wenzhou Medical College, Wenzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weaver CS, Rusyniak DE, Brizendine EJ, Abel S, Somerville GG, Howard JD, Root T. A prospective, randomized, double-blind comparison of buffered versus plain tetracaine in reducing the pain of topical ophthalmic anesthesia. Ann Emerg Med. 2003 Jun;41(6):827-31. doi: 10.1067/mem.2003.192. PMID 12764338
- [Background] Amiel H, Koch PS. Tetracaine hydrochloride 0.5% versus lidocaine 2% jelly as a topical anesthetic agent in cataract surgery: comparative clinical trial. J Cataract Refract Surg. 2007 Jan;33(1):98-100. doi: 10.1016/j.jcrs.2006.09.013. PMID 17189801